CLINICAL TRIAL: NCT04057898
Title: A Phase 2b/3, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, 12 Month Clinical Trial to Evaluate the Efficacy and Safety of MN-166 (Ibudilast) Followed by Open-Label Extension Phase in Subjects With Amyotrophic Lateral Sclerosis
Brief Title: Evaluation of MN-166 (Ibudilast) for 12 Months Followed by an Open-label Extension for 6 Months in Patients With ALS
Acronym: COMBAT-ALS
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: MediciNova (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MN-166-ALS-2301
Record Dates: First submitted 2019-08-06; First posted 2019-08-15 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; MN-166; ibudilast; amyotrophic lateral sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — ibudilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MN-166 (Experimental): Subjects will take MN-166 10 mg capsules, up to 50 mg twice a day for 12 months.
  Interventions: Drug: MN-166
- placebo (Placebo Comparator): Subjects will take up to 5 matching placebo capsules twice a day for 12 months.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: MN-166 — Subjects will take MN-166 for 12 months followed by a 6-month open-label extension phase.
  Other Names: ibudilast
  Arms: MN-166
Drug: placebo — Subjects will take matching placebo for 12 months followed by a 6-month open-label extension phase.
  Arms: placebo

SUMMARY:
A Phase 2b/3 multicenter, randomized, double-blind, placebo-controlled, parallel group study to evaluate the efficacy, safety and tolerability of MN-166 given to ALS participants for 12 months followed by a 6-month open-label extension phase.

DETAILED DESCRIPTION:
This is a Phase 2b/3 multicenter, randomized, double-blind, placebo-controlled, parallel group study to evaluate the efficacy, safety and tolerability of MN-166 followed by an open-label extension phase compared to matching placebo in subjects diagnosed with ALS.

The study will consist of a screening phase (up to 30 days) followed by a double-blind phase (12 months). Following the screening phase, subjects who continue to meet entry criteria will be randomly assigned to one of two treatment groups: MN-166 or matching placebo in a 1:1 ratio. Upon completion of the double-blind phase, subjects will be given the option to continue to the Open-label Extension Phase for a period of six months.

ELIGIBILITY:
Major Inclusion Criteria:

* Male or female subjects age 18 - 80 years, inclusive;
* Diagnosis of familial or sporadic ALS as defined by the El Escorial-Revised (2000) research diagnostic criteria for ALS [clinically definite, clinically probable, probable-laboratory-supported];
* ALS onset of ≤18 months from first clinical signs of weakness prior to screening;
* If currently using riluzole, subject must be on a stable dose for at least 30 days prior to initiation of study drug;
* If currently using edaravone, subject should have completed at least 14 days of their initial treatment cycle prior to initiation of study drug;
* Last documented pulmonary function test result (i.e., slow vital capacity or forced vital capacity) must be greater than or equal to 70% predicted;
* Able to swallow study medication capsules;
* No known allergies to the study drug or its excipients;
* Received pneumococcal vaccine within 6 years prior to starting clinical trial.

Major Exclusion Criteria:

* Confirmed hepatic insufficiency or abnormal liver function (AST and/or ALT >3 times upper limit of normal);
* Currently diagnosed with a clinically significant psychiatric disorder or dementia that would preclude evaluation of symptoms;
* Currently use or treated with parenteral (intramuscular or intravenous) high dose (>25 mg/week) Vitamin B12 within 30 days prior to study drug administration;
* Poor peripheral venous access that will limit the ability to draw blood as judged by the Investigator;
* Currently participating, or has participated in a study with an investigational or marketed compound or device within 30 days or 5 half-lives, whichever is shorter, prior to signing the informed consent;
* Use of tracheostomy or >22/24-hour ventilatory support.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in ALSFRS-R score at Month 12 (or last measurement before death in case of censoring) and survival time. | 12 months
  The amyotrophic lateral sclerosis functional rating scale-revised, or ALSFRS-R, measures the functional status of subjects with ALS. It is based on 12 items, each of which is rated on a 5-point scale (0 to 4). The rate of total functional disability thus ranges from 0 (maximum disability) to 48 (normal function) points.

SECONDARY OUTCOMES:
Mean change from baseline of muscle strength measured by hand-held dynamometry | Baseline, Treatment Phase Week 6, Months 3, 6, 9 and12 time points.
  Hand-held dynamometry, or HHD, is used to measure the force generated by each muscle. The scale ranges from 0 (no visible movement of the part) to 10 (holds test position against strong pressure). Thus, the higher the total score, the higher muscle strength is observed.
Mean change from baseline on quality of life assessed by ALSAQ-5 at Month 12 | 12 months
  The Amyotrophic Lateral Sclerosis Assessment Questionnaire, or ALSAQ-5, is a patient self-report questionnaire specifically designed to measure 5 areas of health: physical mobility, activities of daily living and independence, eating and drinking, communication and emotional functioning. The subject is asked about 5 different areas of difficulties in their daily lives: ability to stand up, use of limbs, consuming solid food, level of speech coherence, and degree of hope about the future.Each question provides 5 choices from which to choose: Never, Rarely, Sometimes, Often, and Always or cannot do at all.
Mean change from baseline of functional activity measured by ALSFRS-R at Month 12 | 12 months
  The ALSFRS-R assessment tool measures the functional status of subjects with ALS. It is based on 12 items, each of which is rated on a 5-point scale (0 to 4). The rate of total functional disability thus ranges from 0 (maximum disability) to 48 (normal function) points. In this context, the ALSFRS-R total score change (lower, same, higher) is documented.
Responders, measured in percent of subjects overall, whose ALSFRS-R total score was stable or improved | 12 months
  Proportion of subjects in which ALSFRS-R total score was stable or improved.
Time to survival | 12 months
  Defined by death or permanent dependency to ventilator or tracheostomy.
Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | 12 months
  The incidence of treatment-emergent adverse events (TEAEs), severity (mild, moderate, severe), as well as relationship to study treatment (not related, possibly related, probably related) and whether they are considered serious.
Changes from Baseline in Laboratory Values | 12 months
  Incidence of out-of-normal-range values and markedly abnormal change from baseline in laboratory safety test variables by treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: Project Management Team, Study Chair — Medicinova Inc
Locations (16):
- United States (10):
  - University of California, Orange, California
  - Mayo Clinic, Jacksonville, Florida
  - Augusta University, Augusta, Georgia
  - Indiana University IU Health Neuroscience Center, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - Hennepin Healthcare Research Institute, Minneapolis, Minnesota
  - SUNY Upstate Medical University, Syracuse, New York
  - Duke University, Durham, North Carolina
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - University of Virginia Health System, Charlottesville, Virginia
- Canada (6):
  - University of Alberta Hospital, Edmonton, Alberta
  - McMaster University Medical Center, Hamilton, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
  - University of Saskatchewan - Sastakoon Hospital, Saskatoon, Saskatchwean
  - Hopital de L'Enfant-Jesus, CHU de Quebec-Universite Laval, Québec

REFERENCES:
- [Derived] Trist BG, Fifita JA, Hogan A, Grima N, Smith B, Troakes C, Vance C, Shaw C, Al-Sarraj S, Blair IP, Double KL. Co-deposition of SOD1, TDP-43 and p62 proteinopathies in ALS: evidence for multifaceted pathways underlying neurodegeneration. Acta Neuropathol Commun. 2022 Aug 25;10(1):122. doi: 10.1186/s40478-022-01421-9. PMID 36008843
- [Derived] Oskarsson B, Maragakis N, Bedlack RS, Goyal N, Meyer JA, Genge A, Bodkin C, Maiser S, Staff N, Zinman L, Olney N, Turnbull J, Brooks BR, Klonowski E, Makhay M, Yasui S, Matsuda K. MN-166 (ibudilast) in amyotrophic lateral sclerosis in a Phase IIb/III study: COMBAT-ALS study design. Neurodegener Dis Manag. 2021 Dec;11(6):431-443. doi: 10.2217/nmt-2021-0042. Epub 2021 Nov 24. PMID 34816762
- See also: This webinar explains the COMBAT-ALS study design and background of MN-166 (ibudilast) as a potential treatment for ALS. — https://youtu.be/dayfOj08_3s